CLINICAL TRIAL: NCT05160935
Title: The Anxiety Level and the Effect on Vital Signs of the Education Given to the Patients Who Will Be Applied Coronary Angiography
Brief Title: Effect of the Education Given to the Patients Who Will Be Applied Coronary Angiography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Sevil PAMUK CEBECİ, Asst.Prof.Dr., Eskisehir Osmangazi University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2021-1
Record Dates: First submitted 2021-11-17; First posted 2021-12-16 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Coronary Angiography; Anxiety; Vital Signs; Education; Nursing; Nursing Care
MeSH Terms: conditions — Anxiety Disorders | interventions — Educational Status

STUDY DESIGN:
Masking Description: Planning the Simple Randomization Method; Since the individuals in the sample group will share the same environment, it is created by separating different days for the experimental group and different days for the control group. It is planned to divide the sample as the control group on odd days and the experimental group on even days. In the selection of both groups, attention will be paid to the similarity of individual characteristics such as age, gender and educational status.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Coronary Angiography Training Manual (Experimental): It is the form prepared by the researchers in line with the literature information and the opinion of the specialist physician was taken. It contains information about coronary artery disease, what to do before coronary angiography procedure and what kind of situations await individuals after the procedure.
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Education — Each patient will be informed about the study, and written consent will be obtained from patients who agree to participate in the study, explaining the purpose and duration of the study. A Patient Identification Form will be filled, the patient's vital signs will be evaluated, and the State-Trait Anxiety Inventory will be administered to the patient.
  Before the coronary angiography procedure, the patients in the experimental group will be trained by the researchers using the training booklet. Trait Anxiety Inventory will be re-administered to the patients after the procedure. Vital signs of patients will be monitored.
  In the control group; In line with the information in the patient consent form before the coronary angiography procedure, verbal information will be given about the coronary angiography procedure within the scope of the routine procedure in the clinic. After the procedure, the State-Trait Anxiety Inventory will be applied again. Vital signs will be taken.

SUMMARY:
This research; The aim of this study was to evaluate the effect of the pre-procedural education given to the patients undergoing coronary angiography on the anxiety level and vital signs of the patients.

DETAILED DESCRIPTION:
Coronary Artery Disease is a vascular disease in the category of atherosclerosis, which is characterized by complete or partial occlusion of the arteries, providing oxygen-rich blood to meet the metabolic needs of the heart. It was shown as the top 10 causes of death worldwide in 2017 by the World Health Organization. According to the 2018 data of the Turkish Statistical Institute (TUIK), it has been reported that 39.7% of the deaths caused by the circulatory system in Turkey are due to heart diseases. Coronary angiography, which is among the diagnostic methods of coronary artery disease; It is the process of evaluating the coronary arteries by making them visible by administering radiopaque material to the femoral, brachial, radial and axillary arteries during cardiac catheterization. One of the basic roles of nursing is to provide education for the recovery of the individual and the maintenance of health. In this context, it is thought that nurses' caring about the role of educator in patient care will contribute to reducing the patient's anxiety.

Research; This study was planned to evaluate the effect of pre-procedural education on patients undergoing coronary angiography on their anxiety level and vital signs.

The research was planned as a quasi-experimental study with pretest-posttest control group design between November 2021 and June 2022. The population of all patients who underwent coronary angiography in the Cardiology Service of Eskişehir City Hospital, the sample was calculated using the G-Powr 3.1 program and it was found appropriate to include 79 people in each group with a 95% CI 90% power. The "Simple Randomization Method" will be used to divide the individuals who agree to participate in the research into the experimental and control groups. Since the individuals in the sample group will share the same environment, the experimental group will be included in data collection on even days and the control group on odd days. A "Diagnostic Form" will be filled in for all patients in the sample, their vital signs will be evaluated, and the "State-Trait Anxiety Inventory" will be administered. For the patients in the experimental group; Before the coronary angiography procedure, training will be given by using the "Training Booklet" prepared by the researchers in line with the literature and the opinion of the specialist physician. After the coronary angiography procedure, the "State-Trait Anxiety Inventory" will be re-administered to the patients and their vital signs will be followed. In the control group; Before the coronary angiography procedure, verbal information will be given for the coronary angiography procedure within the scope of the routine procedure in the clinic, in line with the information in the patient consent form. After the procedure, the State-Trait Anxiety Inventory will be applied again. Vital signs will be monitored. The obtained data will be evaluated with appropriate statistical methods.

As a result of the research, it is thought that the questions of whether the education given to the patients who will undergo coronary angiography have an effect on reducing the anxiety levels of the patients and have a positive effect on the vital signs values will be answered.

Keywords: Coronary angiography, anxiety, vital signs, education, nursing, nursing care

This research; The aim of this study was to evaluate the effect of the pre-procedural education given to the patients undergoing coronary angiography on the anxiety level and vital signs of the patients.

Research Questions;

* Does the training given to the patients who will undergo coronary angiography have an effect on the anxiety level of the patients?
* Does the training given to the patients who will undergo coronary angiography have a positive effect on the vital signs of the patients?

ELIGIBILITY:
Inclusion Criteria:

* Having at least literate education level,
* 18 years old or older,
* No communication problems,
* Does not have mental or psychiatric disease,
* Agreeing to participate in the study voluntarily,
* Individuals who will undergo coronary angiography for the first time.

Exclusion criteria:

* Being illiterate
* Being under the age of 18
* Having any communication problem,
* Having mental or psychiatric disease,
* Not wanting to participate in the study,
* Individuals who have undergone coronary angiography before.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
To accept the hypothesis that "the education given to the patients who will undergo coronary angiography has an effect on reducing the anxiety levels of the patients". | 8 weeks
  "State-Trait Anxiety Inventory" will be applied to the patient in the experimental group before the coronary angiography procedure. Then, coronary angiography information training will be given using the Coronary Angiography Training Guide tool. After the angiography procedure, "State-Trait Anxiety Inventory" will be applied again. State-Trait Anxiety Inventory: The inventory includes two separate scales consisting of a total of forty items (twenty items in each scale). For both scales; 0-19 points (absent), 20-39 points (mild), 40-59 points (moderate), 60-79 points (severe), 80 points and above are considered as very severe panic. Both scales have direct and reversed statements. In the State Anxiety Inventory, there are ten in total (1, 2, 5, 8, 10, 11, 15, 16, 19, 20) and in the Trait Anxiety Inventory seven (21, 26, 27, 30, 33, 36, 39) There are reversed statements.
To accept the hypothesis that "the education given to the patients who will undergo coronary angiography has a positive effect on the blood pressure (mm-Hg) level, one of the vital signs values of the patients". | 8 weeks
  The blood pressure (mm-Hg) of the patient in the experimental group before the coronary angiography procedure will be measured and recorded by the nurse. Afterwards, coronary angiography information training will be given audio-visual using the Coronary Angiography Training Guide tool. The patient will be prepared for the coronary angiography procedure. After the coronary angiography procedure, the patient's blood pressure (mm-Hg) will be measured and recorded by the nurse. Pre- and post-procedure scores will be evaluated using appropriate statistical methods. The blood pressure value that is considered normal is 120/80 mm-Hg, with an upper limit of 139/89 mm-Hg.
To accept the hypothesis that "the education given to the patients who will undergo coronary angiography has a positive effect on the heart rate (beats/min) level, which is one of the vital signs values of the patients". | 8 weeks
  Before the coronary angiography procedure of the patient in the experimental group, the heart rate (beats/min) will be measured and recorded by the nurse. Afterwards, coronary angiography information training will be given as audio-visual using the Coronary Angiography Training Guide tool. The patient will be prepared for the coronary angiography procedure. After the coronary angiography procedure, the patient's heart rate (beats/min) will be measured and recorded by the nurse. Pre- and post-procedure scores will be evaluated with appropriate statistical methods. The normal range of pulse rate; 60-100 beats/min.
To accept the hypothesis that "the education given to the patients who will undergo coronary angiography has a positive effect on the vital signs of the patients, the respiratory rate (respiratory rate/min)". | 8 weeks
  The respiratory rate (respiratory rate/min) of the patient in the experimental group before the coronary angiography procedure will be measured and recorded by the nurse. Later, coronary angiography information training will be given audio-visual using the Coronary Angiography Training Guide tool. The patient will be prepared for the coronary angiography procedure. After the coronary angiography procedure, the patient's respiratory rate (respiratory rate/min) will be measured and recorded by the nurse. Pre- and post-procedure scores will be evaluated using appropriate statistical methods. The normal range of respiratory rate; 12-20 ventilation/min.
To accept the hypothesis that "the education given to the patients who will undergo coronary angiography has a positive effect on the vital signs values of the patients and the body temperature (°C) level". | 8 weeks
  Before the coronary angiography procedure of the patient in the experimental group, the body temperature (°C) will be measured and recorded by the nurse. Afterwards, coronary angiography information training will be given as audio-visual using the Coronary Angiography Training Guide tool. The patient will be prepared for the coronary angiography procedure. After the coronary angiography procedure, the patient's body temperature (°C) will be measured and recorded by the nurse. Pre- and post-procedure scores will be evaluated using appropriate statistical methods. The range of body temperature considered normal; 36°C - 38°C
To accept the hypothesis that "the education given to the patients who will undergo coronary angiography has a positive effect on the oxygen saturation (SpO2) level, one of the vital signs values of the patients". | 8 weeks
  Before the coronary angiography procedure of the patient in the experimental group, the oxygen saturation (SpO2) will be measured and recorded by the nurse. Afterwards, coronary angiography information training will be given as audio-visual using the Coronary Angiography Training Guide tool. The patient will be prepared for the coronary angiography procedure. After the patient's coronary angiography procedure, the oxygen saturation (SpO2) will be measured and recorded by the nurse. Pre- and post-procedure scores will be evaluated using appropriate statistical methods. Oxygen saturation (SpO2) is within the considered normal range; 93-100 SpO2.

CONTACTS AND LOCATIONS:
Overall Officials: Sevil PAMUK CEBECİ, Study Director — sevil.pamukcebeci@ogu.edu.tr
Locations (1):
- Eskişehir Şehir Hastanesi, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No